CLINICAL TRIAL: NCT04513691
Title: A Retrospective Chart Review of Newborns With the Presence of Confirmed or Suspected Maternal Chorioamnionitis and Utilization of the Early Onset Sepsis Calculator
Brief Title: A Chart Review of Newborns With the Presence of Confirmed or Suspected Maternal Chorioamnionitis and Utilization of the Early Onset Sepsis Calculator
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Collaborators: Banner University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 641575377
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-09

CONDITIONS: Maternal; Chorioamnionitis, Affecting Fetus; Early-Onset Sepses, Neonatal
MeSH Terms: conditions — Chorioamnionitis; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sample: Asymptomatic newborns 35 weeks or greater GA born at Banner - University Medical Center Phoenix whose mothers were determined or suspected to have CAM.
  Interventions: Diagnostic Test: EOS Calculator

INTERVENTIONS:
Diagnostic Test: EOS Calculator — Neonatal Early-Onset Sepsis Risk Calculator which is a tool that determines the risk of EOS for a particular newborn by looking at maternal risk factors and the newborn's clinical picture as opposed to just laboratory tests alone

SUMMARY:
This study will review practices in relation to chorioamnionitis (CAM) before and after to the implementation of the Neonatal Early-Onset Sepsis (EOS) Risk Calculator to determine the effect in the nursery at Banner - University Medical Center Phoenix. Newborns enrolled will be at least 35 weeks gestational age (GA) and have a maternal diagnosis of at least suspected or confirmed CAM. The data will include those newborns whose assessment and treatment were not guided by the EOS calculator which was implemented on August 28, 2019 and those with which the EOS calculator was utilized. A secondary objective is to show the economic impact with utilization of the EOS calculator. Data collected will include full laboratory workups including complete blood counts (CBC), blood cultures, antibiotic usage, length of time in the newborn nursery and total length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic newborns 35 weeks or greater GA born at Banner - University Medical Center Phoenix whose mothers were determined or suspected to have CAM.

Exclusion Criteria:

* Direct NICU Admissions
* Subjects may be excluded at Investigator discretion

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asymptomatic newborns 35 weeks or greater GA born at Banner - University Medical Center Phoenix April 28, 2018 through April 28, 2020 whose mothers were determined or suspected to have CAM.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
To determine whether the usage of Neonatal EOS Calculator decreased antibiotic usage in newborns with a maternal diagnosis of suspected or confirmed chorioamnionitis (CAM) in our newborn nursery. | August 28, 2018 through August 28, 2020
  To determine the usage of EOS Calculator measuring decreased antibiotic usage.
To determine whether the usage of Neonatal EOS Calculator measuring laboratory testing in newborns with a maternal diagnosis of suspected or confirmed chorioamnionitis (CAM) in our newborn nursery. | August 28, 2018 through August 28, 2020
  To determine the usage of EOS Calculator measuring laboratory testing.
To determine whether the usage of Neonatal EOS Calculator LOS in newborns with a maternal diagnosis of suspected or confirmed chorioamnionitis (CAM) in our newborn nursery. | August 28, 2018 through August 28, 2020
  To determine the usage of EOS Calculator measuring length of stay (LOS) in newborns

SECONDARY OUTCOMES:
To evaluate the economic impact after the implementation of the EOS Calculator in antibiotic usage in newborn nursery and total length of hospital stay. | August 28, 2018 through August 28, 2020
  Evaluate the economic impact after the implementation of the EOS Calculator in antibiotic usage.
To evaluate the economic impact after the implementation of the EOS Calculator in laboratory tests in newborn nursery and total length of hospital stay. | August 28, 2018 through August 28, 2020
  Evaluate the economic impact after the implementation of the EOS Calculator in laboratory tests.
To evaluate the economic impact after the implementation of the EOS Calculator in LOS in newborn nursery and total length of hospital stay. | August 28, 2018 through August 28, 2020
  Evaluate the economic impact after the implementation of the EOS Calculator LOS in newborn nursery and total length of hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Banner - University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No